CLINICAL TRIAL: NCT06637319
Title: Prevalence of Major Vessels Underlying the Potential Incision Site for Emergency Front of Neck Airway Access in Adult Surgical Patients With Impalpable Neck Anatomy
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0099-E
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-09

CONDITIONS: Airway Complication of Anesthesia
Keywords: font of neck access; blood vessels; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy volunteers > 18 years of age
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan of blood vessels where front of neck access vertical incision would take place in a cant intubate cant oxygenate scenario

SUMMARY:
Patients undergoing general anesthesia require assistance with their breathing and with the delivery of oxygen to their lungs. To achieve this, an anesthesiologist inserts a type of plastic breathing tube into the airway via the mouth called an endotracheal tube or laryngeal mask airway. In rare circumstances, the anesthesiologist may not be able to adequately provide oxygen via these methods. In this life-threatening situation, an anesthesiologist may be forced to make an incision in the front of the neck to access the trachea (windpipe) so that emergency oxygen can be provided. This life-saving technique is known as emergency front-of-neck access (eFONA) and is used to prevent low oxygen levels which cause irreversible brain damage and/or death.

This rarely performed procedure carries a risk of harm from bleeding, injury to the airway or inability to access the trachea to provide oxygen. Emergency front of neck access is more likely to be required in patients with abnormal airway anatomy, for example, in patients with obesity and large neck circumference, neck cancer, or a history of head and neck radiation therapy. Though the optimal technique for eFONA is not clear, prominent guidelines advise the use of an 8-10cm incision upwards from the top of the breastbone in order to identify airway structures which cannot be easily felt by the anesthesiologist from the front of the intact neck. This differs from patients who have airway structures which may be easily located at the front of the neck, whereby a smaller incision may be made or a needle inserted into the trachea (widepipe) to provide oxygen. The neck contains major blood vessels which lie close to the airway and these blood vessels may be injured during the 8-10cm incision, creating further difficulty accessing the airway to provide life-saving oxygen.

This study aims to assess for the presence and size of major blood vessels which may be damaged by this incision by using non-invasive ultrasound which will be placed on the skin of your neck to assess for such blood vessels prior to you undergoing anesthesia.

Our study aims to assess the normal anatomy in the adult population such as yourself to understand what to expect when managing patients who require this life-saving therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Ability to understand the rationale of the study assessments and to provide signed consent
* Ability to safely and comfortably take part in the study protocol

Exclusion Criteria:

* Participant refusal
* Participant less than 18 years old or older than 80 years old
* Participants who do not speak English or cannot give informed written consent without assistance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of blood vessels | During the procedure (30 minutes
  The prevalence of blood vessels at front of neck on ultrasound where an emergency front of neck access vertical incision would take place. In total five regions looked at: sternal notch, thyroid gland, cricoid cartilage, cricothyroid membrane and thyroid cartilage

SECONDARY OUTCOMES:
Depth of blood vessels | During the procedure (10 minutes)
  The height from skin to each blood vessels found on ultrasound
Diameter of blood vessels | During the procedure (10 minutes)
  The widest measured diameter of each blood vessels on ultrasound
Distance from midline | During procedure (10 minutes)
  The distance of each blood vessel from midline on ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No